CLINICAL TRIAL: NCT03070522
Title: Randomized Controlled Trial of Prednisone in Cystic Fibrosis Pulmonary Exacerbations
Brief Title: Prednisone in Cystic Fibrosis Pulmonary Exacerbations
Acronym: PIPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Valerie Waters, Staff physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB1000053825
Record Dates: First submitted 2017-02-08; First posted 2017-03-03 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cystic Fibrosis Pulmonary Exacerbation
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Active Comparator): Placebo
  Interventions: Drug: Placebos
- Treatment (Active Comparator): Prednisone
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — oral prednisone for 7 days during pulmonary exacerbation
  Arms: Treatment
Drug: Placebos — Placebo
  Arms: Placebo

SUMMARY:
This will be a 5 year randomized, double blind, placebo controlled trial of 7 days of oral prednisone in cystic fibrosis (CF) patients receiving intravenous (IV) antibiotic treatment for a pulmonary exacerbation at the Hospital for Sick Children and other study sub-sites across Canada. The intervention will be oral prednisone 2 mg/kg/day (max 60 mg) divided twice daily for 7 days as an adjunctive therapy for pulmonary exacerbations in CF patients who have not recovered their baseline forced expiratory volume in 1 second (FEV1) after 7 days of IV antibiotic treatment. The primary outcome will be the proportion of subjects who achieve >90% of their baseline FEV1 % predicted at day 14 of IV antibiotic treatment for a pulmonary exacerbation in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF by newborn screening or at least one clinical feature of CF, AND either (a) or (b) as follows:
2. A documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis
3. A genotype with two identifiable CF-causing mutations
4. Age > 6 years old.
5. Acute pulmonary exacerbation treated with IV antibiotics as previously defined 10% relative drop in FEV1 from baseline at the time of exacerbation
6. Informed consent by patient or parent/legal guardian
7. Ability to reproducibly perform pulmonary function testing
8. Ability to comply with medication use including the ability to take capsules, study visits and study procedures as judged by the site investigator

Exclusion Criteria:

1. A respiratory tract culture positive for Burkholderia cenocepacia in the 12 months prior to enrollment
2. A respiratory tract culture positive for Mycobacterium abscessus in the 12 months prior to enrollment
3. Treatment with IV or oral corticosteroids within 2 weeks of enrollment or from Day 0-Day 7 of the pulmonary exacerbation
4. Active allergic bronchopulmonary aspergillosis (ABPA) at the time of enrollment as determined by treating physician
5. Asthma related exacerbation at enrollment as defined by the treating physician based on clinically compatible symptoms (eg. wheeze)
6. History of avascular necrosis or pathologic bone fracture
7. Uncontrolled hypertension with end organ damage
8. Active gastrointestinal bleeding
9. Status post lung or other organ transplantation
10. Pregnancy
11. Lactose intolerance (contained in placebo)
12. On Lumacaftor-Ivacaftor (Orkambi) at the time of exacerbation
13. Investigational drug use within 30 days prior to enrollment visit
14. Physical findings that would compromise the safety of the subject or the quality of the study data as determined by site investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-10-07 (Actual); Study Completion 2023-10-07 (Actual)

PRIMARY OUTCOMES:
Lung function recovery | At 14 days of antibiotic therapy
  The proportion of subjects who achieve >90% of their baseline FEV1 % predicted at day 14 of IV antibiotic treatment for a PEx in each treatment arm.

SECONDARY OUTCOMES:
lung function recovery at follow up visit | 1 month follow up
  The proportion of subjects who achieve >90% of their baseline FEV1 % predicted
change in pulmonary function testing | at day 7, 14 and 1 month follow up
  change in pulmonary function testing
quality of life as measured by CFQ-R questionnaire | at day 7, 14 and 1 month follow up
  quality of life
quality of life as measured by CF Respiratory Symptom Diary | at day 7, 14 and 1 month follow up
  quality of life
length of hospitalization | Through study completion, up to 100 weeks
  length of hospitalization
time to subsequent pulmonary exacerbation | 1 year follow up time
  time to subsequent pulmonary exacerbation
number of adverse events | At day day 14 of antibiotic therapy and 1 month follow up
  number of adverse events
change in sputum inflammatory markers | at day 7, 14 and 1 month follow up
  change in sputum inflammatory markers
change in serum inflammatory markers | at day 7, 14 and 1 month follow up
  change in serum inflammatory markers
Duration of antibiotic treatment | Through study completion, up to 100 weeks
  Duration of antibiotic treatment

CONTACTS AND LOCATIONS:
Locations (12):
- Canada (12):
  - The Governers of The University of Calgary - Alberta Health Services, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - London Health Sciences Centre - Lawson Health Research Institute, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Unity Health Toronto - St. Michael's Hospital, Toronto, Ontario
  - SickKids, Toronto, Ontario
  - The Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec
  - University of Saskatchewan - Saskatchewan Health Authority, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Waters V, Shaw M, Perrem L, Quon BS, Tullis E, Solomon M, Rayment JH, Lavoie A, Tse SM, Daigneault P, Bilodeau L, Price A, Nicholson M, Chin M, Parkins M, McKinney ML, Tam JS, Stanojevic S, Grasemann H, Ratjen F; (PIPE Study Investigators). A randomised trial of oral prednisone for cystic fibrosis pulmonary exacerbation treatment. Eur Respir J. 2024 Jun 6;63(6):2302278. doi: 10.1183/13993003.02278-2023. Print 2024 Jun. PMID 38697648

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT03070522/Prot_SAP_000.pdf